CLINICAL TRIAL: NCT01448291
Title: The Effects of the Etonogestrel 0.12mg/Ethinyl Estradiol 0.015mg Vaginal Ring (NuvaRing®) on Vaginal Innate and Inflammatory Biomarkers
Brief Title: Effect of the Etonogestrel 0.12mg/Ethinyl Estradiol 0.015mg Vaginal Ring on Vaginal Innate and Inflammatory Biomarkers
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eastern Virginia Medical School (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Thomas Kimble, Assistant Professor, Eastern Virginia Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRC-NVR11; 11-01-FB-0003 (Other: EVMS IRB)
Record Dates: First submitted 2011-07-08; First posted 2011-10-07 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Vaginosis, Bacterial
Keywords: Contraception; Nuvaring; Vaginal inflammation; Bacterial vaginosis; Nugent score
MeSH Terms: conditions — Vaginosis, Bacterial; Vaginitis | interventions — etonogestrel; NuvaRing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nuvaring (Experimental): This is a single-group study in which data points after use of the etonogestrel/ethinyl estradiol vaginal ring will be compared to baseline.
  Interventions: Drug: Etonogestrel /Ethinyl Estradiol Contraceptive Vaginal Ring

INTERVENTIONS:
Drug: Etonogestrel /Ethinyl Estradiol Contraceptive Vaginal Ring — Etonogestrel 0.12mg/Ethinyl Estradiol 0.015mg Vaginal Ring (NuvaRing®) for 3 months
  Other Names: NuvaRing®

SUMMARY:
It is not known if the use of NuvaRing® alters these innate and inflammatory biomarkers of inflammation.

Hypothesis:

The hypothesis is that NuvaRing® will alter inflammatory biomarkers of inflammation, such as vaginal defensin and cytokine levels, resulting in an overall anti-inflammatory milieu in the vagina.

Specific aims of this study are to:

1. Determine biomarkers of inflammation, including defensins and cytokines, concentrations in women with normal vaginal flora (Nugent Score 0 - 3) before and after NuvaRing® use
2. Determine changes in the integrity of cervicovaginal epithelium and leukocytic concentration before and after treatment with NuvaRing®
3. Monitor for changes in the Nugent score before and after NuvaRing® use
4. Assess the antimicrobial activity of vaginal fluid before and after NuvaRing® use
5. Assess HIV infectivity ex vivo on biopsy specimens before and after NuvaRing® use

Methods This is a prospective, open-label, nonrandomized study. Participants will serve as their own controls. The Clinical Research Center of Eastern Virginia Medical School, Norfolk, Virginia, U.S.A. will be the only study site.

DETAILED DESCRIPTION:
1. To complete specific aim #1, the investigators will use commercially available elisa kits to measure human defensins, inflammatory cytokines, and anti-inflammatory cytokines in vaginal fluid washings collected before and after use of NuvaRing.
2. To complete specific aim #2, the investigators will collect biopsies of the uterine cervix before and after NuvaRing use. Specimens will undergo histopathological measures for overall appearance, epithelial integrity, epithelial thickness, leukocyte infiltration, congestion, and edema. The investigators will quantitate the number of CD45+ and NFkB+ cells using immunohistology in the cervical epithelium.

ELIGIBILITY:
Inclusion Criteria:

1. Women (age 18 - 45) interested in using NuvaRing® for contraception for 3 or more months, and women who are not at risk for pregnancy (i.e. abstinent, tubal sterilization, partner with vasectomy)
2. Women with a normal menstrual cycle (21-35 days) for the past three cycles
3. Women with normal pelvic anatomy (by physical exam)
4. Negative urine pregnancy test
5. Normal pap smear within the past 12 months

Exclusion Criteria:

1. Pregnancy
2. Current breastfeeding
3. Less than 6 weeks post partum
4. Current IUD or Implanon use
5. Depot Medroxyprogesterone Acetate use within the past 6 months
6. Current diagnosis of uterine infection
7. Use of hormonal contraception within the past 30 days
8. Current cervical dysplasia
9. Chronic immune suppression
10. Chronic use of immune suppressors such as steroids
11. Chronic antibiotic use
12. Diabetes or fasting blood glucose >105
13. Hysterectomy
14. Uncontrolled hypertension (systolic BP≥140/ diastolic BP≥ 90)
15. Migraine headaches complicated by aura or focal neurologic deficits
16. Menopause
17. Standard contraindications to combined oral contraceptive use (thrombophilia, active liver disease, active deep venous thrombosis, history of thrombosis)
18. Use of tobacco products ≥ 35 years of age
19. Two or more symptomatic genital herpes simplex virus (HSV) outbreaks in past 12 months
20. Human immunodeficiency virus
21. Vulvovaginal candidiasis
22. Trichamonas vaginalis
23. Neisseria gonorrhea
24. Chlamydia trachomatis
25. Bacterial vaginosis
26. Nugent scores of 4 or greater
27. Use of any other study medication within the past 30 days

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-10 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Determine biomarkers of inflammation, including defensins and cytokines, concentrations in women with normal vaginal flora (Nugent Score 0 - 3) after 3 months of NuvaRing® use | 3 months

SECONDARY OUTCOMES:
Determine changes in the integrity of cervicovaginal epithelium and leukocytic concentration after 3 months of treatment with NuvaRing® | Baseline and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas D Kimble, MD, Principal Investigator — Eastern Virginia Medical School/CONRAD
Locations (1):
- Clinical Research Center at Eastern Virginia Medical School, Norfolk, Virginia, United States

REFERENCES:
- [Background] Iqbal SM, Kaul R. Mucosal innate immunity as a determinant of HIV susceptibility. Am J Reprod Immunol. 2008 Jan;59(1):44-54. doi: 10.1111/j.1600-0897.2007.00563.x. PMID 18154595
- [Background] Valore EV, Park CH, Igreti SL, Ganz T. Antimicrobial components of vaginal fluid. Am J Obstet Gynecol. 2002 Sep;187(3):561-8. doi: 10.1067/mob.2002.125280. PMID 12237628
- [Background] Fan SR, Liu XP, Liao QP. Human defensins and cytokines in vaginal lavage fluid of women with bacterial vaginosis. Int J Gynaecol Obstet. 2008 Oct;103(1):50-4. doi: 10.1016/j.ijgo.2008.05.020. Epub 2008 Jul 16. PMID 18635180
- [Background] John M, Keller MJ, Fam EH, Cheshenko N, Hogarty K, Kasowitz A, Wallenstein S, Carlucci MJ, Tuyama AC, Lu W, Klotman ME, Lehrer RI, Herold BC. Cervicovaginal secretions contribute to innate resistance to herpes simplex virus infection. J Infect Dis. 2005 Nov 15;192(10):1731-40. doi: 10.1086/497168. Epub 2005 Oct 13. PMID 16235171
- [Background] Cherpes TL, Marrazzo JM, Cosentino LA, Meyn LA, Murray PJ, Hillier SL. Hormonal contraceptive use modulates the local inflammatory response to bacterial vaginosis. Sex Transm Infect. 2008 Feb;84(1):57-61. doi: 10.1136/sti.2007.026625. Epub 2007 Oct 2. PMID 17911138